CLINICAL TRIAL: NCT02237079
Title: Bazedoxifene/Conjugated Estrogens (BZA/CE) Improvement of Metabolism (BIM)
Acronym: BIM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tulane University Health Sciences Center (Other)
Responsible Party: Principal Investigator, Franck Mauvais-Jarvis, Professor of Medicine, Tulane University Health Sciences Center
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WI190523
Record Dates: First submitted 2014-08-26; First posted 2014-09-11 (Estimated); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-05

CONDITIONS: Obesity; Glucose Homeostasis; Postmenopausal Symptoms
MeSH Terms: conditions — Obesity | interventions — bazedoxifene; Estrogens, Conjugated (USP)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bazedoxifene/Conjugated Estrogens (BZA/CE) (Experimental): Participants assigned to BZA/CE will receive a daily tablet containing conjugated estrogens 0.45 mg and bazedoxifene 20 mg. BZA/CE (bazedoxifene/conjugated estrogens) tablets, 0.45 mg/20 mg are oval, biconvex, pink tablets, branded with "0.45/20" in black ink on one side. The recommended and only FDA approved dosage is one BZA/CE tablet daily, taken without regard to meals. Tablets should be swallowed whole. If a dose of BZA/CE is missed, participants will be instructed to take it as soon as remembered unless it is almost time for the next scheduled dose. They should not take two doses at the same time. The dose is one tablet per day independent of weight and fat mass. Participants will be provided with information about BZA/CE and its potential side effects and contraindications.
  Interventions: Drug: Bazedoxifene/Conjugated Estrogens (BZA/CE)
- Placebo (Placebo Comparator): Participants assigned to placebo will receive a daily tablet that matches the BZA/CE to maintain the blind. Placebo tablets, 0.45 mg/20 mg are oval, biconvex, pink tablets, branded with "0.45/20" in black ink on one side. Also to assure the blind is maintain, participants in the placebo group will be given the same instructions for taking the study medication.Tablets should be swallowed whole. If a dose, participants will be instructed to take it as soon as remembered unless it is almost time for the next scheduled dose. They should not take two doses at the same time. The dose is one tablet per day independent of weight and fat mass. Participants will be provided with information about BZA/CE and its potential side effects and contraindications, again to maintain the blind.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Bazedoxifene/Conjugated Estrogens (BZA/CE) — Daily tablet containing conjugated estrogens 0.45 mg and bazedoxifene 20 mg.
  Other Names: DUAVEE
  Arms: Bazedoxifene/Conjugated Estrogens (BZA/CE)
Drug: Placebo Oral Tablet — Daily placebo tablet
  Arms: Placebo

SUMMARY:
The goal of this pilot clinical study is to perform a randomized placebo-controlled study to assess the beneficial effect of a 3 month-treatment with Bazedoxifene/Conjugated Estrogens (BZA/CE) vs. placebo on glucose homeostasis and body composition in 20 post-menopausal women. The recruitment will be performed at Tulane Health Sciences Center.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women (<5y since final menstrual period) with age between 50-60y
* Symptomatic (hot flashes, vaginal dryness) or asymptomatic
* BMI 26-45 kg/m2 (Overweight, Obesity I and Obesity II)
* Fasting glucose <125mg/dl
* Triglycerides <200mg/dl
* Normal mammogram within past 12 months
* Physician clearance

Exclusion Criteria:

* Amenorrhea from other causes (Hyperandrogenemia and anovulation)
* type 2 and type 1 diabetes
* Medications: diabetes or diabetic drugs, dyslipidemia, estrogen/progestin therapy, antidepressants and antipsychotics, antiretroviral (HIV), oral steroids, weight loss drugs
* ≤ 3 month washout of birth control pill (often prescribed for postmenopausal symptoms)
* Hysterectomy (partial or complete)
* Contraindications to estrogen treatment (unusual vaginal bleeding, blot clots, hepatic disease, bleeding disorder, past/present history of breast or uterine cancer, pregnant, breastfeeding)

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franck Mauvais-Jarvis, MD, Principal Investigator — Tulane University
Locations (1):
- Tulane University Clinical Translational Unit, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
At this time there is no plan to share individual participant data (IPD)

RESULTS

PARTICIPANT FLOW:
Groups:
- Bazedoxifene/Conjugated Estrogens (CE/BZA): Participants assigned to CE/BZA will receive a daily tablet containing conjugated estrogens 0.45 mg and bazedoxifene 20 mg.
- Placebo: Participants assigned to placebo will receive a daily tablet that matches the CE/BZA to maintain the blind.
Period: Overall Study
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Started | 10 | 7
Completed | 7 | 5
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Conjugated Estrogens/Bazedoxifene (CE/BZA): Participants assigned to CE/BZA will receive a daily tablet containing conjugated estrogens 0.45 mg and bazedoxifene 20 mg.
- Total: Total of all reporting groups
Arm/Group | Conjugated Estrogens/Bazedoxifene (CE/BZA) | Placebo | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 54 [52 to 56] | 55 [54 to 58] | 54.5 [53 to 56.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12
Years since last menstrual period (LMP) [Median (Inter-Quartile Range); unit: Years] | 2 [1.4 to 3.8] | 4.5 [2.1 to 4.8] | 2.7 [1.7 to 4.4]
Waist-to-hip ratio [Median (Inter-Quartile Range); unit: Ratio] | 0.9 [0.82 to 0.95] | 0.84 [0.82 to 0.85] | 0.85 [0.82 to 0.94]
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: Kg/m^2] | 33 [30.6 to 37] | 31.2 [30.7 to 38.6] | 32.4 [30.7 to 37.8]
Waist circumference [Median (Inter-Quartile Range); unit: Cm] | 109.2 [91.4 to 114.3] | 106.7 [92 to 116.8] | 108 [91.7 to 115.6]
Fasting glucose [Median (Inter-Quartile Range); unit: mg/dL] | 94 [83 to 114] | 88 [84 to 98] | 93.5 [83.5 to 108]
Total cholesterol [Median (Inter-Quartile Range); unit: mg/dL] | 208 [167 to 218] | 216 [202 to 245] | 211.5 [190.5 to 231.5]
High-density lipoprotein (HDL) [Median (Inter-Quartile Range); unit: mg/dL] | 60 [45 to 69] | 66 [58 to 73] | 63 [49.5 to 71]
Low-density lipoprotein (LDL) [Median (Inter-Quartile Range); unit: mg/dL] | 120 [99 to 148] | 128 [115 to 147] | 124 [111.5 to 147.5]
Triglycerides [Median (Inter-Quartile Range); unit: mg/dL] | 124 [81 to 131] | 103 [102 to 125] | 113.5 [82.5 to 128.5]

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Mass Index
Description: Body composition will be assessed through change in body mass index at baseline and at 3 months post-treatment.
Time Frame: Change at 3 months from baseline
Measure: Median (Inter-Quartile Range); unit: Kg/m^2
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Number analyzed (Participants) | 7 | 5
Kg/m^2 | -0.2 [-0.5 to 0.3] | -0.5 [-0.6 to -0.3]

2. Primary Outcome: Effect of CE/BZA on Body Composition Using Waist-to-hip Ratio
Description: Body composition will be assessed through change in waist-to-hip ratio at baseline and at 3 months post-treatment.
Time Frame: Change at 3 months from baseline
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Number analyzed (Participants) | 7 | 5
Ratio | -0.05 [-0.06 to 0.03] | 0.00 [-0.02 to 0.00]

3. Primary Outcome: Change in Body Composition Using Dual-energy X-ray Absorptiometry (DXA)
Description: Dual-Energy X-ray Absorptiometry was used to assess body composition. DXA uses an x-ray technique to look at the density of the body and can then estimate the amount of lean muscle mass and fat tissue. Body composition will be assessed through change in DXA body composition at baseline and at 3 months post-treatment.
Time Frame: Change at 3 months from baseline
Measure: Median (Inter-Quartile Range); unit: g
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Number analyzed (Participants) | 7 | 5
g
  Total fat mass | 273 [-571 to 974] | -1408 [-1932 to 467]
  Android fat mass | 1.5 [-226 to 611] | -131 [-452 to -86]
  Gynoid fat mass | -26 [-550 to 279] | -178 [-189 to -116]
  Visceral adipose tissue (VAT) mass | 46 [-63 to 118] | -47 [-134 to -23]

4. Primary Outcome: Change in Acute Insulin Response to Glucose (AIRg)
Description: This will be assessed through an IV Glucose Tolerance Test (IVGTT) conducted at baseline and 3 months to measure the change in acute insulin response to glucose. IVGTT data derived by MINMOD Millennium software. MINMOD: a computer program to calculate insulin sensitivity and pancreatic responsivity from the frequently sampled intravenous glucose tolerance test. Acute Insulin Response (AIRg) to Intravenous Glucose is based on glucose and insulin levels obtained during the frequently sampled intravenous glucose tolerance test and calculated using a mathematical model. AIRg is measured as the magnitude of the insulin response to an intravenous glucose injection following glucose administration. A low AIRg indicates decreased ability of the pancreas to secrete insulin.
Time Frame: Change at 3 months from baseline
Population: Note that for technical reasons, the IVGTT serum was processed in only 11 of 12 subjects (CE/BZA n = 6).
Measure: Median (Inter-Quartile Range); unit: uU/l^-1.min^-1
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Number analyzed (Participants) | 6 | 5
uU/l^-1.min^-1 | 189 [-31 to 444] | -25 [-47 to -9]

5. Primary Outcome: Change in Basal Glucose Concentration (Gb)
Description: This will be assessed through an IV Glucose Tolerance Test (IVGTT) conducted at baseline and 3 months to measure the change in basal glucose concentration. IVGTT data derived by MINMOD Millennium software.
Time Frame: Change at 3 months from baseline
Population: Note that for technical reasons, the IVGTT serum was processed in only 11 of 12 subjects (CE/BZA n = 6).
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Number analyzed (Participants) | 6 | 5
mg/dL | -5.2 [-9.2 to -1.7] | 2.7 [0.9 to 4.9]

6. Primary Outcome: Change in Disposition Index (DI)
Description: Disposition index (DI) is the product of insulin sensitivity times the amount of insulin secreted in response to blood glucose levels. DI is commonly used as a measure of β-cell function. This will be assessed through an IV Glucose Tolerance Test (IVGTT) conducted at baseline and 3 months to measure the change in disposition index (DI). IVGTT data derived by MINMOD Millennium software. DI is based on glucose and insulin levels obtained during the frequently sampled intravenous glucose tolerance test and calculated using a mathematical model. DI is the product of insulin sensitivity and the amount of insulin secreted in response to blood glucose levels. Disposition index is used as a measure of beta cell function and the ability of the body to dispose of a glucose load. A low DI is indicative of a higher risk of developing diabetes.
Time Frame: Change at 3 months from baseline
Population: Note that for technical reasons, the IVGTT serum was processed in only 11 of 12 subjects (CE/BZA n = 6).
Measure: Median (Inter-Quartile Range); unit: Index
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Number analyzed (Participants) | 6 | 5
Index | 500 [-19 to 841] | 267 [28 to 572]

7. Primary Outcome: Change in Insulin Sensitivity (SI) Index
Description: SI indicates the net capacity for insulin to promote the disposal of glucose and to inhibit the endogenous production of glucose. This will be assessed through an IV Glucose Tolerance Test (IVGTT) conducted at baseline and 3 months to measure the change in insulin sensitivity (SI) index. IVGTT data derived by MINMOD Millennium software. SI is based on glucose and insulin levels obtained during the frequently sampled intravenous glucose tolerance test and calculated using a mathematical model. SI is a measure of tissue response to circulating insulin in the blood following glucose injection. A low SI signifies low insulin sensitivity and high SI represents high insulin sensitivity.
Time Frame: Change at 3 months from baseline
Population: Note that for technical reasons, the IVGTT serum was processed in only 11 of 12 subjects (CE/BZA n = 6).
Measure: Median (Inter-Quartile Range); unit: uU/L^-1.min^-1
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Number analyzed (Participants) | 6 | 5
uU/L^-1.min^-1 | -0.24 [-1.50 to 0.19] | 1.35 [1.12 to 1.82]

8. Primary Outcome: Change in Homeostatic Model Assessment (HOMA) β-cell Function
Description: The homeostasis model assessment of β-cell function (HOMA-β) is an index of insulin secretory function derived from fasting plasma glucose and insulin concentrations. This will be assessed at baseline and 3 months to measure the change in Homeostatic model assessment (HOMA) β-cell function. (HOMA) β-cell function is a method used to quantify beta-cell function from fasting blood samples of insulin and glucose. Normal levels for (HOMA) β-cell function is 107 or more. Lower numbers mean higher risk of developing diabetes.
Time Frame: Change at 3 months from baseline
Population: Note that for technical reasons, the IVGTT serum was processed in only 11 of 12 subjects (CE/BZA n = 6).
Measure: Median (Inter-Quartile Range); unit: uU/mM
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Number analyzed (Participants) | 6 | 5
uU/mM | 18.5 [-0.9 to 320.6] | -25.5 [-39.9 to 0.1]

9. Primary Outcome: Change in Homeostatic Model Assessment (HOMA) Insulin Resistance (IR)
Description: Homeostatic model assessment (HOMA) is a method for assessing β-cell function and insulin resistance (IR) from basal (fasting) glucose and insulin or C-peptide concentrations. This will be assessed at baseline and 3 months to measure the change in Homeostatic model assessment (HOMA) insulin resistance. HOMA IR is a method used to quantify insulin resistance from fasting blood samples of insulin and glucose. Normal levels for HOMA-IR is less than 2.0. Higher levels mean higher risk for developing diabetes.
Time Frame: Change at 3 months from baseline
Population: Note that for technical reasons, the IVGTT serum was processed in only 11 of 12 subjects (CE/BZA n = 6).
Measure: Median (Inter-Quartile Range); unit: mM.uU/L^-2
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Number analyzed (Participants) | 6 | 5
mM.uU/L^-2 | 0.15 [-0.18 to 0.34] | -0.01 [-0.10 to 0.24]

10. Primary Outcome: Change in Fasting Insulin Clearance (FIC)
Description: This will be assessed at baseline and 3 months to measure the change in fasting insulin clearance (FIC). FIC derived from fasting C-peptide to insulin ratio.
Time Frame: Change at 3 months from baseline
Population: Note that for technical reasons, the IVGTT serum was processed in only 11 of 12 subjects (CE/BZA n = 6).
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Number analyzed (Participants) | 6 | 5
Ratio | -3.50 [-11.56 to 0.78] | -0.25 [-0.70 to -0.00]

11. Primary Outcome: Change in Glucose-stimulated Insulin Clearance (GSIC)
Description: This will be assessed through an IV Glucose Tolerance Test (IVGTT) conducted at baseline and 3 months to measure the change in glucose-stimulated insulin clearance (GSIC). GSIC derived from molar ratio of C-peptide to insulin area under curve (AUC) over first 20 min of IVGTT.
Time Frame: Change at 3 months from baseline
Population: Note that for technical reasons, the IVGTT serum was processed in only 11 of 12 subjects (CE/BZA n = 6).
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Number analyzed (Participants) | 6 | 5
Ratio | -32.8 [-123.6 to 6.9] | -1.85 [-20.5 to 25.8]

12. Secondary Outcome: Measure Change in Serum Biomarkers Panel 1
Description: Systematic inflammation will be measured through change in serum biomarkers (Leptin, Lipocalin 2 (LCN2), plasminogen activator inhibitor-1 (PAI-1), Intact OCN) taken at baseline and 3 months.
Time Frame: Change at 3 months from baseline
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Number analyzed (Participants) | 7 | 5
ng/mL
  Leptin | -1.6 [-7.2 to 9.5] | 0.7 [-0.1 to 10.5]
  Lipocalin-2 (LCN2) | -1.7 [-3 to 3.5] | -3.8 [-4.9 to 2.2]
  Plasminogen activator inhibitor-1 (PAI-1) | -1.8 [-5.2 to -1.4] | 1.3 [-0.4 to 3.3]
  Osteocalcin (OCN) | 0.8 [-0.7 to 3.1] | -0.9 [-1.1 to 2.7]

13. Secondary Outcome: Measure Change in Serum Biomarkers Panel 2
Description: Systematic inflammation will be measured through change in serum biomarkers (Adiponectin, RBP4) taken at baseline and 3 months.
Time Frame: Change at 3 months from baseline
Measure: Median (Inter-Quartile Range); unit: ug/mL
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Number analyzed (Participants) | 7 | 5
ug/mL
  Retinol binding protein 4 (RBP4) | -0.4 [-5.6 to 14.5] | -4.0 [-24.1 to 4.6]
  Adiponectin | -1.4 [-2.8 to -0.5] | -2.5 [-2.6 to -0.4]

14. Secondary Outcome: Measure Change in Leptin:Adiponectin Ratio (LAR)
Description: Systematic inflammation will be measured through change in leptin:adiponectin ratio (LAR) taken at baseline and 3 months.
Time Frame: Change at 3 months from baseline
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Number analyzed (Participants) | 7 | 5
Ratio | 2.71 [-0.04 to 4.96] | 1.55 [0.02 to 4.03]

15. Secondary Outcome: Measure Change in Fibroblast Growth Factor-21 (FGF-21)
Description: Systematic inflammation will be measured through change in Fibroblast growth factor-21 (FGF-21) taken at baseline and 3 months.
Time Frame: Change at 3 months from baseline
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Number analyzed (Participants) | 7 | 5
pg/mL | -134 [-208 to 24] | -89 [-226 to -48]

16. Secondary Outcome: Measure Change in C-Reactive Protein (CRP)
Description: Systematic inflammation will be measured through change in C-Reactive Protein (CRP) taken at baseline and 3 months.
Time Frame: Change at 3 months from baseline
Measure: Median (Inter-Quartile Range); unit: mg/mL
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Number analyzed (Participants) | 7 | 5
mg/mL | -0.41 [-2.66 to 0.45] | -0.39 [-0.82 to -0.06]

17. Secondary Outcome: Measure Change in Thiobarbituric Acid Reactive Substance (TBARS)
Description: Systematic inflammation will be measured through change in Thiobarbituric acid reactive substance (TBARS) taken at baseline and 3 months.
Time Frame: Change at 3 months from baseline
Measure: Median (Inter-Quartile Range); unit: nmol/mL
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
Number analyzed (Participants) | 7 | 5
nmol/mL | -1.7 [-3.3 to -0.4] | -1.2 [-1.2 to 0.0]

ADVERSE EVENTS:
Time Frame: The data were collected during baseline visit (during IVGTT for 3 hours) and then again they were collected at the 3 months visit (during IVGTT for 3 hours).
Arm/Group | Bazedoxifene/Conjugated Estrogens (CE/BZA) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bazedoxifene/Conjugated Estrogens (CE/BZA) (N=7) | Placebo (N=5)
Lower Insulin dose given (Endocrine disorders) | 0 (0) | 1 (1) — During the preparations for IVGTT, incorrect (lower) weight of the subject was used to calculate insulin dose, therefore patient was given lower than recommended insulin dose during IVGTT. This event did not affect patient's wellbeing or health.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT02237079/Prot_SAP_000.pdf